CLINICAL TRIAL: NCT06918613
Title: Ultrasonographic Evaluation of the Effects of Different Wrist Positions on the Median Nerve in Patients With Generalized Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmet Alkım Özkan, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPRMTRH1A
Record Dates: First submitted 2025-04-01; First posted 2025-04-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hypermobility Syndrome (Disorder); Ultrasonography; Median Nerve
Keywords: Generalized Joint Hypermobility; Median Nerve; Ultrasonography; Wrist Positions; Neural Mobility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Generalized Joint Hypermobility: Subjects in this group are diagnosed with Generalized joint hypermobility. Asymptomatic ( no arthralgia, subluxation, pain etc.) subjects with Beighton score 5 or more are included in this group. Full wrist range of motion is required.
  Ultrasonography of median nerve in proximal carpal tunnel will be done in different wrist positions.
- Healthy: This group consists of healthy volunteers. Full wrist range of motion is required. Beighton scores must be 4 or lower.
  Ultrasonography of median nerve in proximal carpal tunnel will be done in different wrist positions.

SUMMARY:
The aim of this study was to evaluate the effects of different wrist positions (neutral, flexion, extension, and ulnar deviation) on median nerve morphology in patients with generalized joint hypermobility (GJH) using ultrasonography and to compare them with healthy controls.

The investigators' hypothesis is that the deformability of the median nerve in response to active maximal wrist flexion, extension, or ulnar deviation may be increased in patients with GJH

DETAILED DESCRIPTION:
This prospective cross-sectional study will include 18 female patients diagnosed with GJH (Beighton score ≥5) and 18 healthy volunteers with similar age, gender, and body mass index. Both wrists of all participants (total of 72 wrists) will be evaluated using ultrasonography. Images of the median nerve will be obtained in neutral position, active maximal flexion, extension, and ulnar deviation. The cross-sectional area and perimeter of the median nerve will be measured in each position, and circularity will be calculated. Deformation ratios will be determined.

Ultrasonographic Evaluation

Ultrasonographic evaluation was performed using a Mindray DC-7 ultrasound device. The ultrasonographic imaging of participants was performed while the shoulder was in neutral position with the forearm resting on a fixed surface in supination, and with the patient sitting in a chair facing the doctor. Images were obtained from both median nerves of the participants. A linear probe was used for imaging the median nerve. The proximal carpal tunnel was defined as the area between the pisiform and scaphoid tubercle; these two anatomical structures were palpated in the palm and easily identified on ultrasound by their hyperechoic surface and strong posterior acoustic shadowing characteristics. The linear probe was placed along the pisiform and scaphoid bones, the probe was kept perpendicular to the median nerve to prevent anisotropic artifact, and the median nerve was visualized in the proximal carpal tunnel.

The wrists of the participants were imaged for the median nerve in the following positions:

Neutral position (fingers in extension) Active maximal flexion position Active maximal ulnar deviation position Active maximal extension position

During position changes, the probe was kept stable and its position was checked before capturing the image. Images were recorded via the ultrasound device.

To test the consistency of ultrasound measurements, imaging of 10 individuals was performed twice with a one-day interval. Measurements were taken and compared. Intraclass correlation coefficient and intra-observer error values were calculated.

Ultrasound Image Analysis

The "ImageJ" program was used to calculate the perimeter and area of the median nerve. The measurement scale in the ultrasound images was proportioned to the number of pixels on the computer screen. Measurements were repeated 3 times and the average of the values was taken.

The circularity formula was defined. A circularity value of 1 indicates that the drawn polygon is a perfect circle; a value less than 1 indicates a deviation from a circle (for example, an oval or irregularly shaped polygon).

To evaluate the deformability of the median nerve, area, perimeter, and circularity deformation ratios were calculated. The deformation ratio was defined as the normalization of the value in different positions with the value in the neutral position. A deformation ratio close to 1 indicates that the ratio in different positions is very similar to the neutral position. The more the deformation ratio deviates from 1, the greater the difference between parameter measurements in neutral and other positions.

Statistical Analysis

The conformity of the variables in the study to normal distribution was evaluated using the Shapiro-Wilk test. Mean±Standard Deviation and Median (Minimum-Maximum) values were used to display the descriptive statistics of the variables.

For comparing Area, Perimeter, Circularity, Area Deformation Ratio, Perimeter Deformation Ratio, and Circularity Deformation Ratio values according to Patient-Control grouping, Independent Samples T-test was used for parameters showing normal distribution, and Mann-Whitney U test was used for parameters not showing normal distribution.

In examining the relationships between Beighton score, age, height, weight, BMI values and Area, Perimeter, Circularity, Area Deformation Ratio, Perimeter Deformation Ratio, Circularity Deformation Ratio values, Pearson correlation analysis was used for parameters conforming to normal distribution, and Spearman non-parametric correlation coefficient was provided for examining relationships between parameters not conforming to normal distribution.

IBM SPSS Statistics 21.0 (IBM Corp. Released 2012. IBM SPSS Statistics for Windows, Version 21.0. Armonk, NY: IBM Corp.) and MS-Excel 2007 programs were used for statistical analyses and calculations. Statistical significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 15-45 years of age
* Female gender
* Diagnosed with GJH according to the hypermobility spectrum disorders definition
* Patients who agree to participate in the study and provide written consent

Exclusion Criteria:

* Having wrist pain
* Inability to complete full range of motion in the wrist joint
* Patients diagnosed with carpal tunnel syndrome
* Anatomical abnormalities (bifid median nerve, aberrant persistent median artery, Martin-Gruber or other anastomoses)
* History of trauma, operation, fracture, or steroid injection of the hand/wrist
* History of known rheumatological, hereditary, genetic disease, or connective tissue disease other than GJH
* Having neurological disease affecting hand functions (cervical radiculopathy, peripheral nerve lesion, polyneuropathy, cerebrovascular event, etc.)
* Patients with history of regular steroid or non-steroid use, receiving oral glucosamine/hyaluronate supplementation
* Those with systemic diseases (inflammatory joint diseases, diabetes mellitus, acromegaly, hypothyroidism, kidney failure, etc.)
* Having a body mass index (BMI) of 30 or above, or history of morbid obesity
* Being pregnant or in lactation period
* Presence of malignancy

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Subjects who met the criteria were selected from those who presented to Istanbul Physical Medicine Rehabilitation Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Area deformation ratio | On the day one of testing
  To evaluate the deformability of the median nerve, deformation ratios for area (mm²), perimeter (mm), and circularity ( Circularity = 4π (Area / Perimeter²) ) is calculated. The deformation ratio is defined as the measurement in the final position divided by the corresponding measurement in the initial position.
Perimeter deformation ratio | On the day one of testing
  To evaluate the deformability of the median nerve, deformation ratios for area (mm²), perimeter (mm), and circularity ( Circularity = 4π (Area / Perimeter²) ) is calculated. The deformation ratio is defined as the measurement in the final position divided by the corresponding measurement in the initial position.
Circularity deformation ratio | On the day one of testing
  To evaluate the deformability of the median nerve, deformation ratios for area (mm²), perimeter (mm), and circularity ( Circularity = 4π (Area / Perimeter²) ) is calculated. The deformation ratio is defined as the measurement in the final position divided by the corresponding measurement in the initial position.

SECONDARY OUTCOMES:
Area | On the day one of testing
  Ultrasonograpic images of median nerve obtained in different wrist positions. The cross-sectional area (mm²) and perimeter (mm) of the median nerve were measured in each position, and circularity (4π (Area / Perimeter²)) was calculated.
Perimeter | On the day one of testing
  Ultrasonograpic images of median nerve obtained in different wrist positions. The cross-sectional area (mm²) and perimeter (mm) of the median nerve were measured in each position, and circularity (4π (Area / Perimeter²)) was calculated.
Circularity | On the day one of testing
  Ultrasonograpic images of median nerve obtained in different wrist positions. The cross-sectional area (mm²) and perimeter (mm) of the median nerve were measured in each position, and circularity (4π (Area / Perimeter²)) was calculated.
Beighton Score | On the day one of testing
  Correlation between Beighton Score, Height (cm), Weight (kg), BMI (kg/m²) and ultrasonographic measurements is investigated
Height | On the day one of testing
  Correlation between Beighton Score, Height (cm), Weight (kg), BMI (kg/m²) and ultrasonographic measurements is investigated
Weight | On the day one of testing
  Correlation between Beighton Score, Height (cm), Weight (kg), BMI (kg/m²) and ultrasonographic measurements is investigated
BMI correlation | On the day one of testing
  Correlation between Beighton Score, Height (cm), Weight (kg), BMI (kg/m²) and ultrasonographic measurements is investigated

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)

REFERENCES:
- [Result] Castori M, Tinkle B, Levy H, Grahame R, Malfait F, Hakim A. A framework for the classification of joint hypermobility and related conditions. Am J Med Genet C Semin Med Genet. 2017 Mar;175(1):148-157. doi: 10.1002/ajmg.c.31539. Epub 2017 Feb 1. PMID 28145606
- [Result] Aktas I, Ofluoglu D, Albay T. The relationship between benign joint hypermobility syndrome and carpal tunnel syndrome. Clin Rheumatol. 2008 Oct;27(10):1283-7. doi: 10.1007/s10067-008-0909-x. Epub 2008 Jun 5. PMID 18528726
- [Result] Wang Y, Filius A, Zhao C, Passe SM, Thoreson AR, An KN, Amadio PC. Altered median nerve deformation and transverse displacement during wrist movement in patients with carpal tunnel syndrome. Acad Radiol. 2014 Apr;21(4):472-80. doi: 10.1016/j.acra.2013.12.012. PMID 24594417